CLINICAL TRIAL: NCT05891145
Title: The Effect of Remimazolam on Postoperative New-onset Atrial Fibrillation in Patients Undergoing Coronary Artery Bypass Grafting
Brief Title: Remimazolam for Postoperative Atrial Fibrillation
Acronym: RePAF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yangzhou University (Other)
Responsible Party: Principal Investigator, Zhuan Zhang, Director, Yangzhou University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2023-YKL01-16
Record Dates: First submitted 2023-05-17; First posted 2023-06-06 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2023-05

CONDITIONS: Coronary Artery Bypass Grafting; Remimazolam
Keywords: Remimazolam; CABG; Postoperative atrial fibrillation; Postoperative new-onset atrial fibrillation; Coronary artery disease; CAD; Coronary artery bypass graft; Myocardial infarction; Revascularization; Anesthesia; Ischemic heart disease
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Infarction; Myocardial Ischemia | interventions — remimazolam; Midazolam

STUDY DESIGN:
Intervention Model Description: A first open-phase trial in which 50 patients (randomized 1:1 to Remimazolam and control groups) will be enrolled as a pilot study to obtain parameters for sample size calculation. A double-blind randomized controlled trial will be conducted to explore remimazolam's effect on POAF and inflammatory factors' blood levels in patients that receive selective CABG.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: 1. The random numbers will be generated by the Power Analysis and Sample Site Software 9.0 (PASS 9.0), sealed with envelopes, and assigned in the order of enrollment by researchers. The randomized envelopes shall only be opened before anesthesia and resealed right after the operation.
  2. Unblinding of results: the monitoring committee did the data unblinding after all enrollment, follow-up, and data entry. Unblinded data was limited to the data monitoring committee and statistical analysts.
  3. Patients can have emergency unblinding under the following conditions: 1) serious adverse events; 2) The result of the unblinding was needed for the following treatment. 3) other emergency situations that investigators thought necessary for unblinding, the detailed reasons need to be recorded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Remimazolam group (Experimental): General anesthesia was induced with 0.1 mg/kg of remimazolam and maintained with 0.1 mg•kg-1•h-1 remimazolam.
  Interventions: Drug: Remimazolam
- Control group (Active Comparator): General anesthesia was induced with 0.1 mg/kg midazolam.
  Interventions: Drug: midazolam

INTERVENTIONS:
Drug: Remimazolam — Remimazolam is dispensed at 2 mg/ml by the designated researchers who are not involved in enrollment, anesthesia administration, and postoperative follow-up.
  Arms: Remimazolam group
Drug: midazolam — Midazolam is dispensed at 1 mg/ml by the designated researchers who are not involved in enrollment, anesthesia administration, and postoperative follow-up.
  Arms: Control group

SUMMARY:
Atrial fibrillation (AF) is the most common cardiac severe arrhythmia globally and is associated with an increased risk of mortality and morbidity, with a loss of 6.0 million disability-adjusted life-years worldwide in 2017, conferring 0.24% of total disability-adjusted life-years globally. Due to the absence of knowledge of AF pathogenesis, currently, available therapies do not prevent AF onset or progression in 85% of patients. Despite the identification of novel druggable targets that are involved in the pathogenesis of AF, the translation of these findings to clinical drug studies is limited.

Postoperative atrial fibrillation (POAF) is the most common type of secondary AF. The incidence of POAF after coronary artery bypass grafting (CABG) is approximately 30%. About 16% of patients developed POAF in cardiac surgery even with the international guideline recommended perioperative beta-blocker intervention.

Remimazolam is a newly approved benzodiazepine sedative indicated for the induction and maintenance of procedural sedation in adults, with significantly reduced sedation and recovery time. It was also found to be with an anti-inflammatory effect and therefore might have an impact on POAF since AF is closely related to the inflammatory response of myocardial tissue and inflammatory factors such as TNF-α. So, the RePAF trial intends to explore whether remimazolam application in induction and maintenance for general anesthesia during cardiac surgery can reduce the incidence of POAF in patients with CABG, and the effect on the postoperative plasma levels of inflammatory factors and stress factors.

DETAILED DESCRIPTION:
Postoperative atrial fibrillation (POAF) presented a 30% incidence in cardiac surgery and 16% even under beta-blocker treatment, leading to serious complications. Inflammation is a key mechanism that promotes POAF. Remimazolam is a newly approved benzodiazepine sedative with anti-inflammatory effects. However, the impact of remimazolam on POAF remains unknown.

To explore whether or not remimazolam can reduce the POAF in coronary artery bypass grafting (CABG) patients, a first open-phase trial in which 50 patients (randomized 1:1 to Remimazolam and control groups) will be enrolled as a pilot study to obtain parameters for sample size calculation. A double-blind randomized controlled trial will be then conducted to explore remimazolam's effect on POAF and inflammatory factors' blood levels in patients that receive selective CABG.

The blood level of inflammatory factors, stress factors (epinephrine, norepinephrine, cortisol, adrenocorticotropic hormone, corticotropin-releasing hormone), myocardial injury markers, and hemodynamic parameters will also be assessed.

This 2-phase clinical trial will provide novel evidence for the newly approved sedative drug, remimazolam, and with detailed data for inflammatory and myocardial injury endpoints.

ELIGIBILITY:
Inclusion Criteria:

* 50-70 years old;
* BMI 18-28 kg/m2；
* Selective CABG surgery will be performed at the Yangzhou Institute Heart and Great Vessels, the Affiliated Hospital of Yangzhou University, Yangzhou, China.
* Patients agree to participate in this study and sign the informed consent form.

Exclusion Criteria:

* Emergency surgery;
* with any other type of cardiac surgery;
* pre-operative supraventricular arrhythmia;
* with moderate or severe valve disease before surgery;
* with a history of chemotherapy or radiotherapy;
* with a history of thoracic or cardiovascular surgery;
* diuretics usage before the surgery.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
postoperative Atrial Fibrillation (POAF) | 7 days after the operation.
  POAF is defined as postoperative new-onset Atrial Fibrillation (AF) lasting more than the 30 s or hemodynamic instability requiring treatment. AF is defined as 1) irregular R-R interval (in the presence of AV conduction), 2) P-wave disappearance, and 3) irregular atrial activity according to the AHA guidelines.

SECONDARY OUTCOMES:
Inflammatory factors | 1) immediately after the operation, 2) 24 hours after the operation.
  Blood level of TNF-α
Stress factors | 1) immediately after the operation, 2) 24 hours after the operation.
  Blood level of epinephrine, norepinephrine, cortisol, adrenocorticotropic hormone, corticotropin-releasing hormone.

OTHER OUTCOMES:
Myocardial injury markers | 7 days after the operation.
  Myocardial injury markers (cTnT, cTnI, CK-MB)
Arterial blood pressure (BP) | 7 days after the operation.
  Hemodynamic parameters
Cardiac index (CI) | 7 days after the operation.
  Hemodynamic parameters
systemic vascular resistance (SVR) | 7 days after the operation.
  Hemodynamic parameters
stroke volume variation (SVV) | 7 days after the operation.
  Hemodynamic parameters

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Hospital of Yangzhou University., Yangzhou, Jiangsu, China